CLINICAL TRIAL: NCT01751139
Title: An Epidemiological Surveillance Study to Evaluate the Incidence of Dengue in Endemic Regions of Brazil
Brief Title: An Epidemiological Surveillance Study to Evaluate the Incidence of Dengue in Brazil
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Tropical Disease Foundation (Other); Goncalo Moniz Research Center (Other); Evandro Chagas Research Institute, Bio-Manguinhos Technology and Immunology Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 116606
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Dengue
Keywords: Endemic regions; Brazil; Incidence; Surveillance; Dengue
MeSH Terms: conditions — Dengue | interventions — Data Collection

ARMS (1):
- Total Group (Other): Subjects six months of age and older at the time of enrolment, recruited from randomly selected households originating from preselected mapped communities. Preferably the recruitment period occurred outside of the peak dengue transmission season, and continued until each site had reached its foreseen target. The expected period for recruiting the target sample size was approximately three months. Recruitment of replacement subjects was done during the low dengue transmission and the recruitment period depended on the number of subjects that need to be replaced. Enrolled subjects were subjects who either lived in households in study areas with support from the Family Health Physician Program (FHP) or the Larval Index Rapid Assay (LIRA) or with field research experience in the community (preferred) or where a similar system of mapped communities with potential for surveillance existed.
  Interventions: Procedure: Blood sample collection; Other: Data collection

INTERVENTIONS:
Procedure: Blood sample collection — Blood samples will be collected at each study visit (Day 0, Month 6, Month 12, Month 24, Month 36 and Month 48) and any time during the study that dengue is suspected. Samples collected at scheduled visits will be tested for anti-dengue antibodies. Samples collected at visits for dengue suspicion will be tested for dengue infection diagnosis.
Other: Data collection — Diary logs will be issued to all subjects at every visit, except Month 48 (Day 0, Month 6, Month 12, Month 24, and Month 36), as required. Any completed diary logs will be verified, as applicable. Subjects will be given a diary log in the event of the occurrence of a symptom that may be associated with suspected dengue.

SUMMARY:
The purpose of this study is to estimate the incidence of dengue infection in children and adults in geographically distinct locations of Brazil.

DETAILED DESCRIPTION:
The aim of this study is to generate dengue disease burden data including estimates of incidence rates, prevalence data and the clinical presentation of dengue across different age groups.

The study will be conducted in at least three cities: Rio de Janeiro, Salvador, and Manaus. This study will also prepare potential sites for future clinical trials, by setting up the logistics and training staff on site to enroll a cohort of subjects perform dengue surveillance and other study procedures.

Households will be randomly selected from communities where a registry system is implemented. All individuals in the household will be eligible for participating in the study. This study will be sponsored by GSK and co-funded by GSK and Fiocruz. As study sponsor, GSK will delegate some activities to Fiocruz, according to the provisions in their Cooperative Research and Development Agreement (CRADA).

ELIGIBILITY:
Inclusion Criteria:

* Written, signed or thumb-printed informed consent (and assent when applicable) must be obtained from the subject or subject's parent(s)/legally acceptable representative(s) (LAR(s)). If the subject/subject's parent(s)/LAR(s) are illiterate the consent form will be countersigned by a witness.
* Male or female at least 6 months of age at the time of enrollment.
* Subject and/or subject's parent(s)/LAR(s) who the study staff believes can comply with the requirements of the protocol.
* Subject who plans, at the time of enrollment, to remain at same residence/study area during their study participation period).

Exclusion Criteria:

* Child in care.
* Participation (current or planned) in another epidemiological study or in a clinical trial that would conflict with the current study, based on investigator's judgement.
* Terminal illness or severe mental incapacity.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3300 (Actual)
Dates: Start 2014-02-18 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (5):
- Brazil (5):
  - GSK Investigational Site, Manaus, Amazonas
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Natal, Rio Grande do Norte
  - GSK Investigational Site, Campinas, São Paulo
  - GSK Investigational Site, Rio de Janeiro

REFERENCES:
- [Derived] de Aguiar DF, de Barros ENC, Ribeiro GS, Brasil P, Mourao MPG, Luz K, Aoki FH, Freitas ARR, Calvet GA, Oliveira E, Branco BF, Abreu A, Cheuvart B, Guignard A, de Boer M, Duarte AC, Borges MB, de Noronha TG. A prospective, multicentre, cohort study to assess the incidence of dengue illness in households from selected communities in Brazil (2014-2018). Int J Infect Dis. 2021 Jul;108:443-453. doi: 10.1016/j.ijid.2021.04.062. Epub 2021 Apr 21. PMID 33894353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In December 2017, GSK decided to deprioritize the development of the dengue purified inactivated vaccine (DPIV) candidate. This decision was made due to the significant scientific challenges of dengue vaccine development.
Period: Overall Study
Arm/Group | Total Group
Started | 3300
Completed | 1033
Not Completed | 2267
Not completed — Other | 135
Not completed — Sponsor study termination | 1609
Not completed — Lost to Follow-up | 240
Not completed — Withdrawal by Subject | 251
Not completed — Adverse Event | 1
Not completed — Death | 31

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the According-to-Protocol cohort that included all evaluable subjects who met all eligibility criteria, complying with the procedures defined in the protocol and who had seroprevalence status at first visit of the first year.
Arm/Group | Total Group
Number analyzed (Participants) | 3264
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (20.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1972
  Male | 1292
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate (Per 1000 Person-years) of All Laboratory-confirmed Symptomatic Dengue Infection by Calendar Year
Description: Incidence rate (IR) of laboratory-confirmed symptomatic dengue infection (lab-conf.) with 95% Confidence Interval (CI) for each year and overall, calculated as the incidence rate per 1000 person-years : numerator = number of all lab-conf. cases reported during the follow-up (FU) period at risk; denominator = total Person-years at risk, i.e. sum of FU periods at risk expressed in years until first Reverse Transcriptase quantitative Polymerase Chain Reaction (RT-qPCR) confirmed symptomatic dengue infection or subject's withdrawal, whichever came first. Lab-conf. case defined as follows: Dengue virus identification through RT-qPCR on acute serum sample or Dengue virus NS1 positive on acute serum sample through Enzyme-linked Immunosorbent Assay (ELISA) or Anti-Dengue Immunoglobulin type M (IgM) seroconversion between acute and convalescent serum samples through ELISA. Data were not analyzed by Dengue season as planned in the protocol as most of the cases occurred outside the seasons.
Time Frame: At each calendar year i.e. Year 2014, 2015, 2016, 2017, 2018, and overall calendar years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: infections per 1000 person-year
Arm/Group | Total Group
Number analyzed (Participants) | 3264
infections per 1000 person-year
  Year 2014: number analyzed (Participants) | 1192
  Year 2014 | 1.778 [0.045 to 9.904]
  Year 2015: number analyzed (Participants) | 1823
  Year 2015 | 5.083 [1.865 to 11.063]
  Year 2016: number analyzed (Participants) | 2343
  Year 2016 | 7.428 [4.061 to 12.463]
  Year 2017: number analyzed (Participants) | 2924
  Year 2017 | 5.785 [3.163 to 9.707]
  Year 2018: number analyzed (Participants) | 2804
  Year 2018 | 7.079 [3.962 to 11.676]
  Overall calendar years | 6.123 [4.544 to 8.072]

2. Secondary Outcome: Incidence Rate (Per 1000 Person-years) of All Virologically-confirmed Symptomatic Dengue Infection by Calendar Year
Description: Incidence rate (IR) of virologically-confirmed symptomatic dengue infection with 95% Confidence Interval (CI) for each year separately and overall years calculated as the incidence rate per 1000 person-years : the numerator is the number of all virologically-confirmed dengue infection cases reported during the follow-up period at risk; the denominator is the total Person-years at risk, i.e. sum of the follow-up periods at risk expressed in years. A virologically confirmed symptomatic dengue infection is defined as a dengue case confirmed by RT-qPCR. Data were not analyzed by Dengue season as planned in the protocol as most of the cases occurred outside the seasons. Analysis was not performed by DENV-type as data would not be reliable due to the low number of cases reported.
Time Frame: At each calendar year i.e. Year 2014, 2015, 2016, 2017, 2018, and overall calendar years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: infections per 1000 person-year
Arm/Group | Total Group
Number analyzed (Participants) | 3264
infections per 1000 person-year
  Year 2014: number analyzed (Participants) | 1192
  Year 2014 | 0.000 [0.000 to 6.558]
  Year 2015: number analyzed (Participants) | 1823
  Year 2015 | 2.541 [0.524 to 7.427]
  Year 2016: number analyzed (Participants) | 2343
  Year 2016 | 0.531 [0.013 to 2.956]
  Year 2017: number analyzed (Participants) | 2924
  Year 2017 | 0.413 [0.010 to 2.302]
  Year 2018: number analyzed (Participants) | 2804
  Year 2018 | 1.888 [0.514 to 4.833]
  Overall calendar years | 1.102 [0.504 to 2.092]

3. Secondary Outcome: Incidence Rate (Per 1000 Person-years) of All Laboratory-confirmed or Probable Symptomatic Dengue Infection by Study Site, and Calendar Year
Description: Incidence rate (IR) of laboratory-confirmed or probable symptomatic dengue infection with 95% Confidence Interval (CI) by study site, and for each year separately and overall years calculated as the incidence rate per 1000 person-years : the numerator is the number of all laboratory-confirmed or probable symptomatic dengue infection cases reported during the follow-up period at risk; the denominator is the total Person-years at risk, i.e. sum of the follow-up periods at risk expressed in years. For early presenters, a probable case was that case without laboratory confirmation, presenting IgG positive in the convalescent sample; for late presenters, a probable case was the case without seroconversion of IgM, presenting at least one IgG positive in one sample (acute or convalescent). Data were not analyzed by Dengue season as planned in the protocol as most of the cases occurred outside the seasons.
Time Frame: At each calendar year i.e. Year 2014, 2015, 2016, 2017, 2018, and overall calendar years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: infections per 1000 person-year
Arm/Group | Total Group
Number analyzed (Participants) | 3264
infections per 1000 person-year
  Rio at year 2014: number analyzed (Participants) | 595
  Rio at year 2014 | 18.284 [9.632 to 34.708]
  Rio at year 2015: number analyzed (Participants) | 691
  Rio at year 2015 | 25.666 [17.644 to 37.337]
  Rio at year 2016: number analyzed (Participants) | 592
  Rio at year 2016 | 27.263 [19.592 to 37.938]
  Rio at year 2017: number analyzed (Participants) | 545
  Rio at year 2017 | 17.704 [12.340 to 25.400]
  Rio at year 2018: number analyzed (Participants) | 506
  Rio at year 2018 | 12.761 [8.493 to 19.175]
  Rio overall calendar years: number analyzed (Participants) | 737
  Rio overall calendar years | 19.597 [14.781 to 25.982]
  Manaus at year 2014: number analyzed (Participants) | 597
  Manaus at year 2014 | 27.098 [13.954 to 52.622]
  Manaus at year 2015: number analyzed (Participants) | 597
  Manaus at year 2015 | 38.039 [27.330 to 52.944]
  Manaus at year 2016: number analyzed (Participants) | 549
  Manaus at year 2016 | 40.405 [30.203 to 54.054]
  Manaus at year 2017: number analyzed (Participants) | 634
  Manaus at year 2017 | 26.239 [19.013 to 36.210]
  Manaus at year 2018: number analyzed (Participants) | 598
  Manaus at year 2018 | 18.913 [13.135 to 27.232]
  Manaus overall calendar years: number analyzed (Participants) | 727
  Manaus overall calendar years | 29.044 [22.622 to 37.289]
  Salvador at year 2015: number analyzed (Participants) | 535
  Salvador at year 2015 | 77.398 [52.617 to 113.850]
  Salvador at year 2016: number analyzed (Participants) | 604
  Salvador at year 2016 | 82.213 [65.162 to 103.725]
  Salvador at year 2017: number analyzed (Participants) | 561
  Salvador at year 2017 | 53.388 [40.722 to 69.995]
  Salvador at year 2018: number analyzed (Participants) | 525
  Salvador at year 2018 | 38.482 [27.823 to 53.224]
  Salvador overall calendar years: number analyzed (Participants) | 605
  Salvador overall calendar years | 59.097 [46.242 to 75.525]
  Natal at year 2016: number analyzed (Participants) | 598
  Natal at year 2016 | 71.873 [51.198 to 100.896]
  Natal at year 2017: number analyzed (Participants) | 587
  Natal at year 2017 | 46.674 [34.829 to 62.546]
  Natal at year 2018: number analyzed (Participants) | 582
  Natal at year 2018 | 33.642 [24.002 to 47.154]
  Natal overall calendar years: number analyzed (Participants) | 598
  Natal overall calendar years | 51.664 [37.852 to 70.516]
  Campinas at year 2017: number analyzed (Participants) | 597
  Campinas at year 2017 | 1.688 [0.234 to 12.152]
  Campinas at year 2018: number analyzed (Participants) | 593
  Campinas at year 2018 | 1.217 [0.171 to 8.670]
  Campinas overall calendar years: number analyzed (Participants) | 597
  Campinas overall calendar years | 1.869 [0.260 to 13.429]
  All study sites at year 2014: number analyzed (Participants) | 1192
  All study sites at year 2014 | 18.715 [8.748 to 40.034]
  All study sites at year 2015: number analyzed (Participants) | 1823
  All study sites at year 2015 | 26.271 [15.779 to 43.738]
  All study sites at year 2016: number analyzed (Participants) | 2343
  All study sites at year 2016 | 27.905 [17.883 to 43.543]
  All study sites at year 2017: number analyzed (Participants) | 2924
  All study sites at year 2017 | 18.121 [11.609 to 28.286]
  All study sites at year 2018: number analyzed (Participants) | 2804
  All study sites at year 2018 | 13.061 [8.214 to 20.771]
  All study sites overall calendar years | 20.059 [13.152 to 30.591]

4. Secondary Outcome: Incidence Rate (Per 1000 Person-years) of All Laboratory-confirmed or Probable Symptomatic Dengue Infection by Age Category, and Calendar Year
Description: Incidence rate (IR) of laboratory-confirmed or probable symptomatic dengue infection with 95% Confidence Interval (CI) by age category, and for each year separately and overall years calculated as the incidence rate per 1000 person-years : the numerator is the number of all laboratory-confirmed or probable symptomatic dengue infection cases reported during the follow-up period at risk; the denominator is the total Person-years at risk, i.e. sum of the follow-up periods at risk expressed in years. For early presenters, a probable case was that case without laboratory confirmation, presenting IgG positive in the convalescent sample; for late presenters, a probable case was the case without seroconversion of IgM, presenting at least one IgG positive in one sample (acute or convalescent). Data were not analyzed by Dengue season as planned in the protocol as most of the cases occurred outside the seasons.
Time Frame: At each calendar year i.e. Year 2014, 2015, 2016, 2017, 2018, and overall calendar years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: infections per 1000 person-year
Arm/Group | Total Group
Number analyzed (Participants) | 3264
infections per 1000 person-year
  ≤17 years at year 2014: number analyzed (Participants) | 175
  ≤17 years at year 2014 | 11.826 [0.299 to 65.890]
  ≤17 years at year 2015: number analyzed (Participants) | 442
  ≤17 years at year 2015 | 25.038 [8.130 to 58.429]
  ≤17 years at year 2016: number analyzed (Participants) | 623
  ≤17 years at year 2016 | 47.415 [30.057 to 71.146]
  ≤17 years at year 2017: number analyzed (Participants) | 890
  ≤17 years at year 2017 | 28.345 [17.065 to 44.264]
  ≤17 years at year 2018: number analyzed (Participants) | 866
  ≤17 years at year 2018 | 32.151 [19.902 to 49.147]
  ≤17 years overall calendar years: number analyzed (Participants) | 964
  ≤17 years overall calendar years | 32.970 [25.653 to 41.725]
  18-49 years at year 2014: number analyzed (Participants) | 654
  18-49 years at year 2014 | 9.658 [1.992 to 28.224]
  18-49 years at year 2015: number analyzed (Participants) | 947
  18-49 years at year 2015 | 41.479 [27.095 to 60.776]
  18-49 years at year 2016: number analyzed (Participants) | 1188
  18-49 years at year 2016 | 61.410 [46.748 to 79.215]
  18-49 years at year 2017: number analyzed (Participants) | 1409
  18-49 years at year 2017 | 46.497 [35.123 to 60.380]
  18-49 years at year 2018: number analyzed (Participants) | 1335
  18-49 years at year 2018 | 28.574 [19.136 to 41.037]
  18-49 years overall calendar years: number analyzed (Participants) | 1602
  18-49 years overall calendar years | 42.016 [35.988 to 48.764]
  ≥ 50 years at year 2014: number analyzed (Participants) | 363
  ≥ 50 years at year 2014 | 35.853 [13.157 to 78.037]
  ≥ 50 years at year 2015: number analyzed (Participants) | 434
  ≥ 50 years at year 2015 | 33.908 [17.521 to 59.230]
  ≥ 50 years at year 2016: number analyzed (Participants) | 532
  ≥ 50 years at year 2016 | 50.123 [31.412 to 75.887]
  ≥ 50 years at year 2017: number analyzed (Participants) | 625
  ≥ 50 years at year 2017 | 22.011 [11.373 to 38.448]
  ≥ 50 years at year 2018: number analyzed (Participants) | 603
  ≥ 50 years at year 2018 | 11.091 [3.601 to 25.882]
  ≥ 50 years overall calendar years: number analyzed (Participants) | 698
  ≥ 50 years overall calendar years | 29.138 [22.069 to 37.752]

5. Secondary Outcome: Incidence Rate (Per 1000 Person-years) of All Laboratory-confirmed or Probable Symptomatic Dengue Infection by Gender, and Calendar Year
Description: Incidence rate (IR) of laboratory-confirmed or probable symptomatic dengue infection with 95% Confidence Interval (CI) by gender, and for each year separately and overall years calculated as the incidence rate per 1000 person-years : the numerator is the number of all laboratory-confirmed or probable symptomatic dengue infection cases reported during the follow-up period at risk; the denominator is the total Person-years at risk, i.e. sum of the follow-up periods at risk expressed in years. For early presenters, a probable case was that case without laboratory confirmation, presenting IgG positive in the convalescent sample; for late presenters, a probable case was the case without seroconversion of IgM, presenting at least one IgG positive in one sample (acute or convalescent). Data were not analyzed by Dengue season as planned in the protocol as most of the cases occurred outside the seasons.
Time Frame: At each calendar year i.e. Year 2014, 2015, 2016, 2017, 2018, and overall calendar years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: infections per 1000 person-year
Arm/Group | Total Group
Number analyzed (Participants) | 3264
infections per 1000 person-year
  Female at year 2014: number analyzed (Participants) | 745
  Female at year 2014 | 14.266 [4.632 to 33.291]
  Female at year 2015: number analyzed (Participants) | 1107
  Female at year 2015 | 37.839 [25.144 to 54.688]
  Female at year 2016: number analyzed (Participants) | 1444
  Female at year 2016 | 61.579 [48.094 to 77.674]
  Female at year 2017: number analyzed (Participants) | 1768
  Female at year 2017 | 40.564 [30.954 to 52.214]
  Female at year 2018: number analyzed (Participants) | 1699
  Female at year 2018 | 29.601 [20.948 to 40.630]
  Female overall calendar years: number analyzed (Participants) | 1972
  Female overall calendar years | 40.349 [34.976 to 46.313]
  Male at year 2014: number analyzed (Participants) | 447
  Male at year 2014 | 23.579 [7.656 to 55.026]
  Male at year 2015: number analyzed (Participants) | 716
  Male at year 2015 | 34.056 [19.061 to 56.170]
  Male at year 2016: number analyzed (Participants) | 899
  Male at year 2016 | 45.097 [31.043 to 63.333]
  Male at year 2017: number analyzed (Participants) | 1156
  Male at year 2017 | 28.701 [18.914 to 41.758]
  Male at year 2018: number analyzed (Participants) | 1105
  Male at year 2018 | 20.355 [11.857 to 32.590]
  Male overall calendar years: number analyzed (Participants) | 1292
  Male overall calendar years | 30.694 [24.891 to 37.445]

6. Secondary Outcome: Number of Primary Symptomatic Dengue Infection Cases Among Laboratory-confirmed or Probable Cases
Description: A primary symptomatic dengue case is a subject with laboratory confirmed or probable symptomatic dengue infection, and without evidence of previous dengue infection (absence of Ig G antibodies at the previous scheduled visit and absence of laboratory confirmed symptomatic case detected previously at study surveillance). Analysis was not performed by DENV-type as data would not be reliable due to the low number of cases reported.
Time Frame: From Year 2014 to Year 2018 (a range of 1 to 4 years for an individual subject)
Population: Analysis was performed on the laboratory confirmed or probable symptomatic dengue cases, excluding those reported without fever or reported before the first visit in the first year.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 299
Participants
  Primary symptomatic cases in Rio: number analyzed (Participants) | 53
  Primary symptomatic cases in Rio | 2
  Primary symptomatic cases in Manaus: number analyzed (Participants) | 77
  Primary symptomatic cases in Manaus | 5
  Primary symptomatic cases in Salvador: number analyzed (Participants) | 109
  Primary symptomatic cases in Salvador | 1
  Primary symptomatic cases in Natal: number analyzed (Participants) | 59
  Primary symptomatic cases in Natal | 4
  Primary symptomatic cases in Campinas: number analyzed (Participants) | 1
  Primary symptomatic cases in Campinas | 0
  Overall primary symptomatic cases | 12

7. Secondary Outcome: Number of Secondary Symptomatic Dengue Infection Cases Among Laboratory-confirmed or Probable Cases
Description: A secondary symptomatic dengue case is a subject with laboratory confirmed or probable symptomatic dengue infection, and with evidence of previous dengue infection (presence of IgG antibodies at the previous scheduled visit(s) or laboratory-confirmed symptomatic case detected previously at study surveillance). Analysis was not performed by DENV-type as data would not be reliable due to the low number of cases reported.
Time Frame: From Year 2014 to Year 2018 (a range of 1 to 4 years for an individual subject)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 299
Participants
  Secondary symptomatic cases in Rio: number analyzed (Participants) | 53
  Secondary symptomatic cases in Rio | 51
  Secondary symptomatic cases in Manaus: number analyzed (Participants) | 77
  Secondary symptomatic cases in Manaus | 72
  Secondary symptomatic cases in Salvador: number analyzed (Participants) | 109
  Secondary symptomatic cases in Salvador | 108
  Secondary symptomatic cases in Natal: number analyzed (Participants) | 59
  Secondary symptomatic cases in Natal | 55
  Secondary symptomatic cases in Campinas: number analyzed (Participants) | 1
  Secondary symptomatic cases in Campinas | 1
  Overall secondary symptomatic cases | 287

8. Secondary Outcome: Number of Subjects With Previous Dengue Infection (Dengue Seroprevalence) at Baseline, by Study Site and Overall
Description: A subject was considered as having previous dengue infection at baseline, based on seroprevalence at first visit, namely if Dengue IgG positive (i.e. reactive) at first visit or if Laboratory-confirmed symptomatic dengue case detected at first visit (baseline).
Time Frame: At the first visit of the first year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 3264
Participants
  Seroprevalence at visit 1 in Rio: number analyzed (Participants) | 737
  Seroprevalence at visit 1 in Rio | 604
  Seroprevalence at visit 1 in Manaus: number analyzed (Participants) | 727
  Seroprevalence at visit 1 in Manaus | 583
  Seroprevalence at visit 1 in Salvador: number analyzed (Participants) | 605
  Seroprevalence at visit 1 in Salvador | 580
  Seroprevalence at visit 1 in Natal: number analyzed (Participants) | 598
  Seroprevalence at visit 1 in Natal | 534
  Seroprevalence at visit 1 in Campinas: number analyzed (Participants) | 597
  Seroprevalence at visit 1 in Campinas | 186
  Overall seroprevalence at visit 1 | 2487

9. Secondary Outcome: Number of Subjects With Previous Dengue Infection (Dengue Seroprevalence) at Baseline, by Gender
Description: as for outcome 8
Time Frame: At the first visit of the first year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 3264
Participants
  Seroprevalence at visit 1 in Rio-females: number analyzed (Participants) | 440
  Seroprevalence at visit 1 in Rio-females | 372
  Seroprevalence at visit 1 in Manaus-females: number analyzed (Participants) | 452
  Seroprevalence at visit 1 in Manaus-females | 381
  Seroprevalence at visit 1 in Salvador-females: number analyzed (Participants) | 355
  Seroprevalence at visit 1 in Salvador-females | 341
  Seroprevalence at visit 1 in Natal-females: number analyzed (Participants) | 375
  Seroprevalence at visit 1 in Natal-females | 350
  Seroprevalence at visit 1 in Campinas-females: number analyzed (Participants) | 350
  Seroprevalence at visit 1 in Campinas-females | 112
  Overall seroprevalence at visit 1-females: number analyzed (Participants) | 1972
  Overall seroprevalence at visit 1-females | 1556
  Seroprevalence at visit 1 in Rio-males: number analyzed (Participants) | 297
  Seroprevalence at visit 1 in Rio-males | 232
  Seroprevalence at visit 1 in Manaus-males: number analyzed (Participants) | 275
  Seroprevalence at visit 1 in Manaus-males | 202
  Seroprevalence at visit 1 in Salvador-males: number analyzed (Participants) | 250
  Seroprevalence at visit 1 in Salvador-males | 239
  Seroprevalence at visit 1 in Natal-males: number analyzed (Participants) | 223
  Seroprevalence at visit 1 in Natal-males | 184
  Seroprevalence at visit 1 in Campinas-males: number analyzed (Participants) | 247
  Seroprevalence at visit 1 in Campinas-males | 74
  Overall seroprevalence at visit 1-males: number analyzed (Participants) | 1292
  Overall seroprevalence at visit 1-males | 931

10. Secondary Outcome: Number of Subjects With Previous Dengue Infection (Dengue Seroprevalence) at Baseline, by Age Group at Enrolment
Description: as for outcome 8
Time Frame: At the first visit of the first year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 3264
Participants
  First seroprevalence at ≤17 years in Rio: number analyzed (Participants) | 211
  First seroprevalence at ≤17 years in Rio | 95
  First seroprevalence at ≤17 years in Manaus: number analyzed (Participants) | 203
  First seroprevalence at ≤17 years in Manaus | 85
  First seroprevalence at ≤17 years in Salvador: number analyzed (Participants) | 192
  First seroprevalence at ≤17 years in Salvador | 171
  First seroprevalence at ≤17 years in Natal: number analyzed (Participants) | 178
  First seroprevalence at ≤17 years in Natal | 117
  First seroprevalence at ≤17 years in Campinas: number analyzed (Participants) | 180
  First seroprevalence at ≤17 years in Campinas | 22
  Overall first seroprevalence at ≤17 years: number analyzed (Participants) | 964
  Overall first seroprevalence at ≤17 years | 490
  First seroprevalence at 18-49 years in Rio: number analyzed (Participants) | 358
  First seroprevalence at 18-49 years in Rio | 344
  First seroprevalence at 18-49 years in Manaus: number analyzed (Participants) | 329
  First seroprevalence at 18-49 years in Manaus | 304
  First seroprevalence at 18-49 years in Salvador: number analyzed (Participants) | 324
  First seroprevalence at 18-49 years in Salvador | 320
  First seroprevalence at 18-49 years in Natal: number analyzed (Participants) | 300
  First seroprevalence at 18-49 years in Natal | 297
  First seroprevalence at 18-49 years in Campinas: number analyzed (Participants) | 291
  First seroprevalence at 18-49 years in Campinas | 121
  Overall first seroprevalence at 18-49 years: number analyzed (Participants) | 1602
  Overall first seroprevalence at 18-49 years | 1386
  First seroprevalence at ≥50 years in Rio: number analyzed (Participants) | 168
  First seroprevalence at ≥50 years in Rio | 165
  First seroprevalence at ≥50 years in Manaus: number analyzed (Participants) | 195
  First seroprevalence at ≥50 years in Manaus | 194
  First seroprevalence at ≥50 years in Salvador: number analyzed (Participants) | 89
  First seroprevalence at ≥50 years in Salvador | 89
  First seroprevalence at ≥50 years in Natal: number analyzed (Participants) | 120
  First seroprevalence at ≥50 years in Natal | 120
  First seroprevalence at ≥50 years in Campinas: number analyzed (Participants) | 126
  First seroprevalence at ≥50 years in Campinas | 43
  Overall first seroprevalence at ≥50 years: number analyzed (Participants) | 698
  Overall first seroprevalence at ≥50 years | 611

11. Secondary Outcome: Incidence Rate (Per 1000 Person-years) of Primary Inapparent Dengue Infection by Study Site and Calendar Year, and Overall, Among Subjects With no Seroprevalence at the First Visit
Description: Incidence rate (IR) of primary inapparent dengue infection with 95% Confidence Interval (CI) by site and, for each year separately and overall years calculated as the incidence rate per 1000 person-years, among subjects with no seroprevalence at the first visit: the numerator is the number of all primary inapparent dengue infection cases reported during the follow-up period at risk. The denominator is the total Person-years at risk, i.e. sum of the follow-up periods at risk expressed in years. The primary inapparent dengue infection condition was defined as a documented seroconversion (anti-dengue IgG antibodies) between two sequential sera samples obtained during the scheduled visits without clinical suspicion of dengue (identified during the time period in which seroconversion occurred). Data were not analyzed by Dengue season as planned in the protocol as most of the cases occurred outside the seasons.
Time Frame: At each calendar year i.e. Year 2014, 2015, 2016, 2017, 2018, and overall calendar years
Population: Analysis was performed on the According-to-Protocol cohort that included all evaluable subjects who met all eligibility criteria, complying with the procedures defined in the protocol and who had no seroprevalence at first visit of the first year.
Measure: Number (95% Confidence Interval); unit: infections per 1000 person-year
Arm/Group | Total Group
Number analyzed (Participants) | 777
infections per 1000 person-year
  Primary inapparent dengue in Rio at year 2014: number analyzed (Participants) | 62
  Primary inapparent dengue in Rio at year 2014 | 0.000 [0.000 to 99.997]
  Primary inapparent dengue in Rio at year 2015: number analyzed (Participants) | 129
  Primary inapparent dengue in Rio at year 2015 | 16.570 [0.420 to 92.322]
  Primary inapparent dengue in Rio at year 2016: number analyzed (Participants) | 114
  Primary inapparent dengue in Rio at year 2016 | 48.757 [15.831 to 113.782]
  Primary inapparent dengue in Rio at year 2017: number analyzed (Participants) | 98
  Primary inapparent dengue in Rio at year 2017 | 57.491 [18.667 to 134.165]
  Primary inapparent dengue in Rio at year 2018: number analyzed (Participants) | 89
  Primary inapparent dengue in Rio at year 2018 | 38.610 [4.676 to 139.473]
  Overall primary inapparent dengue in Rio: number analyzed (Participants) | 133
  Overall primary inapparent dengue in Rio | 38.398 [20.445 to 65.662]
  Primary inapparent dengue in Manuas at year 2014: number analyzed (Participants) | 57
  Primary inapparent dengue in Manuas at year 2014 | 0.000 [0.000 to 196.845]
  Primary inapparent dengue in Manuas at year 2015: number analyzed (Participants) | 57
  Primary inapparent dengue in Manuas at year 2015 | 132.246 [48.532 to 287.844]
  Primary inapparent dengue in Manuas at year 2016: number analyzed (Participants) | 47
  Primary inapparent dengue in Manuas at year 2016 | 108.548 [29.576 to 277.926]
  Primary inapparent dengue in Manuas at year 2017: number analyzed (Participants) | 125
  Primary inapparent dengue in Manuas at year 2017 | 19.956 [0.505 to 111.188]
  Primary inapparent dengue in Manuas at year 2018: number analyzed (Participants) | 125
  Primary inapparent dengue in Manuas at year 2018 | 109.613 [52.564 to 201.582]
  Overall primary inapparent dengue in Manuas: number analyzed (Participants) | 144
  Overall primary inapparent dengue in Manuas | 86.673 [53.652 to 132.489]
  Primary inapparent dengue in Salvador at year 2015: number analyzed (Participants) | 19
  Primary inapparent dengue in Salvador at year 2015 | 0.000 [0.000 to 1603.861]
  Primary inapparent dengue in Salvador at year 2016: number analyzed (Participants) | 25
  Primary inapparent dengue in Salvador at year 2016 | 251.256 [81.582 to 586.348]
  Primary inapparent dengue in Salvador at year 2017: number analyzed (Participants) | 23
  Primary inapparent dengue in Salvador at year 2017 | 0.000 [0.000 to 216.230]
  Primary inapparent dengue in Salvador at year 2018: number analyzed (Participants) | 22
  Primary inapparent dengue in Salvador at year 2018 | 0.000 [0.000 to 291.842]
  Overall primary inapparent dengue in Salvador: number analyzed (Participants) | 25
  Overall primary inapparent dengue in Salvador | 96.339 [31.281 to 224.823]
  Primary inapparent dengue in Natal at year 2016: number analyzed (Participants) | 64
  Primary inapparent dengue in Natal at year 2016 | 0.000 [0.000 to 174.415]
  Primary inapparent dengue in Natal at year 2017: number analyzed (Participants) | 62
  Primary inapparent dengue in Natal at year 2017 | 32.648 [3.954 to 117.935]
  Primary inapparent dengue in Natal at year 2018: number analyzed (Participants) | 61
  Primary inapparent dengue in Natal at year 2018 | 150.667 [60.576 to 310.432]
  Overall primary inapparent dengue in Natal: number analyzed (Participants) | 64
  Overall primary inapparent dengue in Natal | 69.838 [31.934 to 132.574]
  Primary inapparent dengue in Campinas at year 2017: number analyzed (Participants) | 411
  Primary inapparent dengue in Campinas at year 2017 | 0.000 [0.000 to 21.600]
  Primary inapparent dengue in Campinas at year 2018: number analyzed (Participants) | 410
  Primary inapparent dengue in Campinas at year 2018 | 12.661 [3.450 to 32.416]
  Overall primary inapparent dengue in Campinas: number analyzed (Participants) | 411
  Overall primary inapparent dengue in Campinas | 8.218 [2.239 to 21.042]
  Overall primary inapparent dengue in 2014: number analyzed (Participants) | 119
  Overall primary inapparent dengue in 2014 | 0.000 [0.000 to 66.323]
  Overall primary inapparent dengue in 2015: number analyzed (Participants) | 205
  Overall primary inapparent dengue in 2015 | 64.803 [26.054 to 133.519]
  Overall primary inapparent dengue in 2016: number analyzed (Participants) | 250
  Overall primary inapparent dengue in 2016 | 77.584 [42.416 to 130.172]
  Overall primary inapparent dengue in 2017: number analyzed (Participants) | 719
  Overall primary inapparent dengue in 2017 | 20.716 [8.944 to 40.818]
  Overall primary inapparent dengue in 2018: number analyzed (Participants) | 707
  Overall primary inapparent dengue in 2018 | 44.396 [28.143 to 66.615]
  Overall primary inapparent dengue overall years | 41.655 [31.110 to 54.625]

12. Secondary Outcome: Incidence Rate (Per 1000 Person-years) of Primary Inapparent Dengue Infection by Age Category and Calendar Year, and Overall, Among Subjects With no Seroprevalence at the First Visit
Description: Incidence rate (IR) of primary inapparent dengue infection with 95% Confidence Interval (CI) by age category and, for each year separately and overall years calculated as the incidence rate per 1000 person-years, among subjects with no seroprevalence at the first visit: the numerator is the number of all primary inapparent dengue infection cases reported during the follow-up period at risk. The denominator is the total Person-years at risk, i.e. sum of the follow-up periods at risk expressed in years. The primary inapparent dengue infection condition was defined as a documented seroconversion (anti-dengue IgG antibodies) between two sequential sera samples obtained during the scheduled visits without clinical suspicion of dengue (identified during the time period in which seroconversion occurred). Data were not analyzed by Dengue season as planned in the protocol as most of the cases occurred outside the seasons.
Time Frame: At each calendar year i.e. Year 2014, 2015, 2016, 2017, 2018, and overall calendar years
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: infections per 1000 person-year
Arm/Group | Total Group
Number analyzed (Participants) | 777
infections per 1000 person-year
  Primary inapparent dengue at ≤17 years in 2014: number analyzed (Participants) | 78
  Primary inapparent dengue at ≤17 years in 2014 | 0.000 [0.000 to 99.565]
  Primary inapparent dengue at ≤17 years in 2015: number analyzed (Participants) | 160
  Primary inapparent dengue at ≤17 years in 2015 | 37.712 [7.777 to 110.211]
  Primary inapparent dengue at ≤17 years in 2016: number analyzed (Participants) | 215
  Primary inapparent dengue at ≤17 years in 2016 | 51.004 [22.020 to 100.498]
  Primary inapparent dengue at ≤17 years in 2017: number analyzed (Participants) | 437
  Primary inapparent dengue at ≤17 years in 2017 | 19.266 [6.255 to 44.959]
  Primary inapparent dengue at ≤17 years in 2018: number analyzed (Participants) | 428
  Primary inapparent dengue at ≤17 years in 2018 | 64.460 [39.374 to 99.553]
  Overall primary inapparent dengue at ≤17 years: number analyzed (Participants) | 474
  Overall primary inapparent dengue at ≤17 years | 42.692 [29.901 to 59.104]
  Primary inapparent dengue at 18-49 years in 2014: number analyzed (Participants) | 37
  Primary inapparent dengue at 18-49 years in 2014 | 0.000 [0.000 to 226.034]
  Primary inapparent dengue at 18-49 years in 2015: number analyzed (Participants) | 41
  Primary inapparent dengue at 18-49 years in 2015 | 160.064 [43.612 to 409.827]
  Primary inapparent dengue at 18-49 years in 2016: number analyzed (Participants) | 32
  Primary inapparent dengue at 18-49 years in 2016 | 291.262 [106.888 to 633.955]
  Primary inapparent dengue at 18-49 years in 2017: number analyzed (Participants) | 196
  Primary inapparent dengue at 18-49 years in 2017 | 22.873 [2.770 to 82.625]
  Primary inapparent dengue at 18-49 years in 2018: number analyzed (Participants) | 194
  Primary inapparent dengue at 18-49 years in 2018 | 14.092 [1.707 to 50.907]
  Overall primary inapparent dengue at 18-49 years: number analyzed (Participants) | 216
  Overall primary inapparent dengue at 18-49 years | 48.065 [26.278 to 80.646]
  Primary inapparent dengue at ≥ 50 years in 2014: number analyzed (Participants) | 4
  Primary inapparent dengue at ≥ 50 years in 2014 | 0.000 [0.000 to 1639.502]
  Primary inapparent dengue at ≥ 50 years in 2015: number analyzed (Participants) | 4
  Primary inapparent dengue at ≥ 50 years in 2015 | 0.000 [0.000 to 1063.078]
  Primary inapparent dengue at ≥ 50 years in 2016: number analyzed (Participants) | 3
  Primary inapparent dengue at ≥ 50 years in 2016 | 0.000 [0.000 to 1225.541]
  Primary inapparent dengue at ≥ 50 years in 2017: number analyzed (Participants) | 86
  Primary inapparent dengue at ≥ 50 years in 2017 | 25.504 [0.646 to 142.098]
  Primary inapparent dengue at ≥ 50 years in 2018: number analyzed (Participants) | 85
  Primary inapparent dengue at ≥ 50 years in 2018 | 15.179 [0.384 to 84.573]
  Overall primary inapparent dengue at ≥ 50 years: number analyzed (Participants) | 87
  Overall primary inapparent dengue at ≥ 50 years | 17.570 [2.128 to 63.469]

13. Secondary Outcome: Incidence Rate (Per 1000 Person-years) of Primary Inapparent Dengue Infection by Gender and Calendar Year, and Overall, Among Subjects With no Seroprevalence at the First Visit
Description: Incidence rate (IR) of primary inapparent dengue infection with 95% Confidence Interval (CI) by gender and, for each year separately and overall years calculated as the incidence rate per 1000 person-years, among subjects with no seroprevalence at the first visit: the numerator is the number of all primary inapparent dengue infection cases reported during the follow-up period at risk. The denominator is the total Person-years at risk, i.e. sum of the follow-up periods at risk expressed in years. The primary inapparent dengue infection condition was defined as a documented seroconversion (anti-dengue IgG antibodies) between two sequential sera samples obtained during the scheduled visits without clinical suspicion of dengue (identified during the time period in which seroconversion occurred). Data were not analyzed by Dengue season as planned in the protocol as most of the cases occurred outside the seasons.
Time Frame: At each calendar year i.e. Year 2014, 2015, 2016, 2017, 2018, and overall calendar years
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: infections per 1000 person-year
Arm/Group | Total Group
Number analyzed (Participants) | 777
infections per 1000 person-year
  Primary inapparent dengue at year 2014- females: number analyzed (Participants) | 58
  Primary inapparent dengue at year 2014- females | 0.000 [0.000 to 129.027]
  Primary inapparent dengue at year 2015- females: number analyzed (Participants) | 102
  Primary inapparent dengue at year 2015- females | 36.792 [4.456 to 132.904]
  Primary inapparent dengue at year 2016- females: number analyzed (Participants) | 119
  Primary inapparent dengue at year 2016- females | 91.002 [39.288 to 179.311]
  Primary inapparent dengue at year 2017- females: number analyzed (Participants) | 385
  Primary inapparent dengue at year 2017- females | 25.219 [8.189 to 58.854]
  Primary inapparent dengue at year 2018- females: number analyzed (Participants) | 377
  Primary inapparent dengue at year 2018- females | 43.176 [22.310 to 75.420]
  Overall Primary inapparent dengue- females: number analyzed (Participants) | 416
  Overall Primary inapparent dengue- females | 41.728 [27.499 to 60.712]
  Primary inapparent dengue at year 2014- males: number analyzed (Participants) | 61
  Primary inapparent dengue at year 2014- males | 0.000 [0.000 to 136.423]
  Primary inapparent dengue at year 2015- males: number analyzed (Participants) | 103
  Primary inapparent dengue at year 2015- males | 93.179 [30.255 to 217.449]
  Primary inapparent dengue at year 2016- males: number analyzed (Participants) | 131
  Primary inapparent dengue at year 2016- males | 64.837 [23.794 to 141.122]
  Primary inapparent dengue at year 2017- males: number analyzed (Participants) | 334
  Primary inapparent dengue at year 2017- males | 15.965 [3.292 to 46.657]
  Primary inapparent dengue at year 2018- males: number analyzed (Participants) | 330
  Primary inapparent dengue at year 2018- males | 45.807 [22.866 to 81.961]
  Overall primary inapparent dengue- males: number analyzed (Participants) | 361
  Overall primary inapparent dengue- males | 41.577 [26.907 to 61.376]

14. Secondary Outcome: Number of Suspected Dengue Cases With Severity Criteria
Description: To describe symptoms and spectrum of dengue disease in the study population for the suspected dengue cases, excluding those reported without fever. Suspected symptomatic dengue case= Febrile illness with body temperature ≥ 38°C measured (by any route) on at least two consecutive days and less than 14 days with or without the presence of other dengue symptoms or signs, without an obvious aetiology unrelated to dengue, based on investigator's judgement; Lab-confirmed = laboratory-confirmed symptomatic dengue cases; Probable = probable symptomatic dengue cases; Negative = negative symptomatic dengue cases; Indeterminate = indeterminate symptomatic dengue case( not classified as laboratory confirmed case, probable case or negative case); Severe dengue episode = at least one criteria met for severe dengue (in accordance to the "dengue with warning signs" and "severe dengue" definitions in the 2009 WHO guidelines for dengue).
Time Frame: From Year 2014 to Year 2018 (a range of 1 to 4 years for an individual subject)
Population: Analysis was performed on the According-to-Protocol cohort that included all evaluable subjects who met all eligibility criteria, complying with the procedures defined in the protocol and who were defined as suspected dengue cases, excluding those without fever or reported before the first visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 1284
Participants
  Severe dengue episode- indeterminate: number analyzed (Participants) | 247
  Severe dengue episode- indeterminate | 0
  Severe dengue episode- lab-confirmed: number analyzed (Participants) | 50
  Severe dengue episode- lab-confirmed | 0
  Severe dengue episode- negative: number analyzed (Participants) | 738
  Severe dengue episode- negative | 0
  Severe dengue episode- probable: number analyzed (Participants) | 249
  Severe dengue episode- probable | 1
  Severe dengue episode- total | 1
  Severe plasma leakage- indeterminate: number analyzed (Participants) | 247
  Severe plasma leakage- indeterminate | 0
  Severe plasma leakage- lab-confirmed: number analyzed (Participants) | 50
  Severe plasma leakage- lab-confirmed | 0
  Severe plasma leakage- negative: number analyzed (Participants) | 738
  Severe plasma leakage- negative | 0
  Severe plasma leakage- probable: number analyzed (Participants) | 249
  Severe plasma leakage- probable | 0
  Severe plasma leakage- total | 0
  Fluid accumulation- indeterminate: number analyzed (Participants) | 247
  Fluid accumulation- indeterminate | 0
  Fluid accumulation- lab-confirmed: number analyzed (Participants) | 50
  Fluid accumulation- lab-confirmed | 0
  Fluid accumulation- negative: number analyzed (Participants) | 738
  Fluid accumulation- negative | 0
  Fluid accumulation- probable: number analyzed (Participants) | 249
  Fluid accumulation- probable | 0
  Fluid accumulation- total | 0
  Severe bleeding- indeterminate: number analyzed (Participants) | 247
  Severe bleeding- indeterminate | 0
  Severe bleeding- lab-confirmed: number analyzed (Participants) | 50
  Severe bleeding- lab-confirmed | 0
  Severe bleeding- negative: number analyzed (Participants) | 738
  Severe bleeding- negative | 0
  Severe bleeding- probable: number analyzed (Participants) | 249
  Severe bleeding- probable | 1
  Severe bleeding- total | 1
  Liver involvement- indeterminate: number analyzed (Participants) | 247
  Liver involvement- indeterminate | 0
  Liver involvement- lab-confirmed: number analyzed (Participants) | 50
  Liver involvement- lab-confirmed | 0
  Liver involvement- negative: number analyzed (Participants) | 738
  Liver involvement- negative | 0
  Liver involvement- probable: number analyzed (Participants) | 249
  Liver involvement- probable | 0
  Liver involvement- total | 0
  Central Nervous System involvement- indeterminate: number analyzed (Participants) | 247
  Central Nervous System involvement- indeterminate | 0
  Central Nervous System involvement- lab-confirmed: number analyzed (Participants) | 50
  Central Nervous System involvement- lab-confirmed | 0
  Central Nervous System involvement- negative: number analyzed (Participants) | 738
  Central Nervous System involvement- negative | 0
  Central Nervous System involvement- probable: number analyzed (Participants) | 249
  Central Nervous System involvement- probable | 0
  Central Nervous System involvement- total | 0
  Heart and other organs involvement- indeterminate: number analyzed (Participants) | 247
  Heart and other organs involvement- indeterminate | 0
  Heart and other organs involvement- lab-confirmed: number analyzed (Participants) | 50
  Heart and other organs involvement- lab-confirmed | 0
  Heart and other organs involvement- negative: number analyzed (Participants) | 738
  Heart and other organs involvement- negative | 0
  Heart and other organs involvement- probable: number analyzed (Participants) | 249
  Heart and other organs involvement- probable | 0
  Heart and other organs involvement- total | 0

15. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Related to a Study Procedure
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Year 2014 to Year 2018 (a range of 1 to 4 years for an individual subject)
Population: Analysis was performed on the Total cohort that included all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 3300
Participants | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events related to study procedure were collected from Year 2014 to Year 2018 (a range of 1 to 4 years for an individual subject).
Description: Other adverse events were not collected in this study.
Arm/Group | Total Group
All-Cause Mortality (participants affected / at risk) | 31/3300
Serious Adverse Events (participants affected / at risk) | 0/3300
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT01751139/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT01751139/SAP_001.pdf